CLINICAL TRIAL: NCT00589537
Title: Trial of Imaging and Schedule in Seminoma Testis
Brief Title: Magnetic Resonance Imaging and Computed Tomography in Patients With Stage I Seminoma of the Testicle
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical Research Council (Other Government)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Diagnostic
Other Study IDs: MRC-NCRI-TRISST-TE24; CDR0000574037 (Registry Identifier: PDQ (Physician Data Query)); EU-20771; ISRCTN65987321
Record Dates: First submitted 2007-12-25; First posted 2008-01-09 (Estimated); Last update posted 2013-08-07 (Estimated); Status verified 2009-07

CONDITIONS: Testicular Germ Cell Tumor
Keywords: testicular seminoma; stage I malignant testicular germ cell tumor
MeSH Terms: conditions — Testicular Germ Cell Tumor; Seminoma; Testicular Neoplasms | interventions — Magnetic Resonance Spectroscopy

INTERVENTIONS:
Other: questionnaire administration
Procedure: computed tomography
Procedure: magnetic resonance imaging
Procedure: quality-of-life assessment

SUMMARY:
RATIONALE: Imaging procedures, such as MRI and CT scan, may find recurrent cancer. It is not yet known which MRI or CT scan schedule is more effective in finding recurrent cancer.

PURPOSE: This randomized phase III trial is comparing four different MRI and CT scan schedules in patients with stage I seminoma of the testicle.

DETAILED DESCRIPTION:
OBJECTIVES:

* To assess whether a reduced computed tomography (CT) schedule or magnetic resonance imaging (MRI) could be used as safe and effective alternatives to standard CT-based surveillance in the management of patients with stage I seminoma of the testis.

OUTLINE: This is a multicenter study. Patients are randomized to 1 of 4 surveillance arms.

* Arm I: Patients undergo computed tomography (CT) scan of the abdomen/retroperitoneum* at 6, 12, 18, 24, 36, 48, and 60 months in the absence of disease progression.
* Arm II: Patients undergo CT scan of the abdomen/retroperitoneum* at 6, 18, and 36 months in the absence of disease progression.
* Arm III: Patients undergo magnetic resonance imaging (MRI) of the abdomen/retroperitoneum* at 6, 12, 18, 24, 36, 48, and 60 months in the absence of disease progression.
* Arm IV: Patients undergo MRI of the abdomen/retroperitoneum* at 6, 18, and 36 months in the absence of disease progression.

NOTE: *Patients with a history of ipsilateral inguino-scrotal surgery also undergo imaging of the pelvis.

Patients complete questionnaires at baseline and periodically during study to assess health-related quality of life; utilization and cost of healthcare services (including the cost of CT- or MRI-based surveillance and the management of any recurrence); and acceptability of allocated scanning schedule.

Patients are followed every 3 months for 2 years, every 4 months for 1 year, and then every 6 months for 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed seminoma of the testis

  * Stage I disease, as determined by clinical examination and CT scan of the chest, abdomen, and pelvis
* No evidence of any non-seminoma germ cell tumor elements
* Has undergone orchidectomy within the past 8 weeks

  * Normal serum alpha-fetoprotein pre-orchidectomy and at study randomization
  * Normal serum beta human chorionic gonadotrophin at study randomization (may have been elevated pre-orchidectomy)
* Not planning to undergo adjuvant therapy

PATIENT CHARACTERISTICS:

* Able to attend regular surveillance
* No other malignancy within the past 10 years expect successfully treated nonmelanoma skin cancer
* No contraindication to MRI (i.e., ferrous metal implants of any type, cardiac pacemaker or defibrillator, or history of injury by metal fragments)

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Min Age: 16 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 660 (Estimated)
Dates: Start 2008-03; Primary Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients relapsing with Royal Marsden Hospital stage IIC or greater disease

SECONDARY OUTCOMES:
Difference in mean abdominal mass size at relapse between computed tomography (CT) scan and magnetic resonance imaging (MRI)
Time on surveillance before detection of relapse
Prospective identification of first modality to detect relapse (patient symptom, clinical examination, tumor marker, chest x-ray, cross-sectional image)
Extent of relapse according to International Germ Cell Cancer Collaborative Group classification
Disease-free survival
Overall survival
Prospective evaluation of prognostic factors for relapse
Number of false positive MRIs
Resource use and costs

CONTACTS AND LOCATIONS:
Overall Officials: Johnathan Joffe, MD, Study Chair — Huddersfield Royal Infirmary
Locations (29):
- United Kingdom (29):
  - Royal Bournemouth Hospital, Bournemouth, England
  - Sussex Cancer Centre at Royal Sussex County Hospital, Brighton, England
  - Bristol Haematology and Oncology Centre, Bristol, England
  - Addenbrooke's Hospital, Cambridge, England
  - Gloucestershire Oncology Centre at Cheltenham General Hospital, Cheltenham, England
  - Huddersfield Royal Infirmary, Huddersfield, West Yorks, England
  - Leeds Cancer Centre at St. James's University Hospital, Leeds, England
  - Leicester Royal Infirmary, Leicester, England
  - Lincoln County Hospital, Lincoln, England
  - UCL Cancer Institute, London, England
  - Charing Cross Hospital, London, England
  - University College of London Hospitals, London, England
  - Mid Kent Oncology Centre at Maidstone Hospital, Maidstone, England
  - Christie Hospital, Manchester, England
  - James Cook University Hospital, Middlesbrough, England
  - Northern Centre for Cancer Treatment at Newcastle General Hospital, Newcastle upon Tyne, England
  - Northampton General Hospital, Northampton, England
  - Mount Vernon Cancer Centre at Mount Vernon Hospital, Northwood, England
  - Nottingham City Hospital, Nottingham, England
  - Churchill Hospital, Oxford, England
  - Berkshire Cancer Centre at Royal Berkshire Hospital, Reading, England
  - Cancer Research Centre at Weston Park Hospital, Sheffield, England
  - Royal Marsden - Surrey, Sutton, England
  - Yeovil District Hospital, Yeovil, England
  - Centre for Cancer Research and Cell Biology at Queen's University Belfast, Belfast, Northern Ireland
  - Aberdeen Royal Infirmary, Aberdeen, Scotland
  - Beatson West of Scotland Cancer Centre, Glasgow, Scotland
  - Velindre Cancer Center at Velindre Hospital, Cardiff, Wales
  - Glan Clwyd Hospital, Rhyl, Denbighshire, Wales

REFERENCES:
- [Derived] Joffe JK, Cafferty FH, Murphy L, Rustin GJS, Sohaib SA, Gabe R, Stenning SP, James E, Noor D, Wade S, Schiavone F, Swift S, Dunwoodie E, Hall M, Sharma A, Braybrooke J, Shamash J, Logue J, Taylor HH, Hennig I, White J, Rudman S, Worlding J, Bloomfield D, Faust G, Glen H, Jones R, Seckl M, MacDonald G, Sreenivasan T, Kumar S, Protheroe A, Venkitaraman R, Mazhar D, Coyle V, Highley M, Geldart T, Laing R, Kaplan RS, Huddart RA; TRISST Trial Management Group and Investigators. Imaging Modality and Frequency in Surveillance of Stage I Seminoma Testicular Cancer: Results From a Randomized, Phase III, Noninferiority Trial (TRISST). J Clin Oncol. 2022 Aug 1;40(22):2468-2478. doi: 10.1200/JCO.21.01199. Epub 2022 Mar 17. PMID 35298280